CLINICAL TRIAL: NCT03877588
Title: Perioperative Nutritional and Hemodinamic Support in Retroperitoneal Sarcoma Patients. A Phase II Prospective Feasibility Study.
Brief Title: Nutritional Status in Retroperitoneal Sarcoma.
Acronym: NOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: INT-91/16
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Retroperitoneal Sarcoma; Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Nutritional Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary retroperitoneal sarcoma (Other): All eligible patients are screened in preoperative phase, at least 30 days before surgery, for presence of protein energetic malnutrition (PEM). PEM is defined according to biochemical and physiological parameters (Table). 3 class of PEM are identified: no PEM, mild PEM and serious PEM. Different nutritional oral supplements are provided according to the degree of malnutrition.
  Interventions: Dietary Supplement: Oral Nutritional Support

INTERVENTIONS:
Dietary Supplement: Oral Nutritional Support — Preoperative oral nutritional support is provided according to malnutrition grade

SUMMARY:
Prospective feasibility study of perioperative nutrition in patients affected by primary retroperitoneal sarcoma

DETAILED DESCRIPTION:
Aim of our study was to investigate the feasibility of a prehabilitation policy to optimize protein energetic reserves in a group of patients affected by primary localized RPS, candidate to a multiple organ resection surgery, as well as the feasibility of a standardized nutritional postoperative caloric target and its adequacy.

ELIGIBILITY:
Inclusion Criteria:

- every patient with retroperitoneal sarcoma scheduled for surgery

Exclusion Criteria:

* chronic renal failure
* diabetes mellitus
* emergency surgery
* physical status classification system ASA>3
* any contraindication to arterial catheter in Femoral artery for PICCO hemodynamic monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of Adherence to protocol | 15 days
  Rate of adherence to prescribed oral nutritional support

REFERENCES:
- [Derived] Previtali P, Fiore M, Colombo J, Arendar I, Fumagalli L, Pizzocri M, Colombo C, Rampello NN, Mariani L, Gronchi A, Codazzi D. Malnutrition and Perioperative Nutritional Support in Retroperitoneal Sarcoma Patients: Results from a Prospective Study. Ann Surg Oncol. 2020 Jun;27(6):2025-2032. doi: 10.1245/s10434-019-08121-0. Epub 2019 Dec 17. PMID 31848820